CLINICAL TRIAL: NCT03117270
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II Study to Assess the Efficacy and Safety of Filgotinib Administered for 12 Weeks to Subjects With Active Ankylosing Spondylitis
Brief Title: A Study to Assess Efficacy and Safety of Filgotinib in Ankylosing Spondylitis
Acronym: TORTUGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-223
Record Dates: First submitted 2017-03-30; First posted 2017-04-17 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral filgotinib tablets (Experimental)
  Interventions: Drug: filgotinib
- placebo tablets (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: filgotinib — one filgotinib oral tablet q.d.
  Arms: oral filgotinib tablets
Drug: Placebo Oral Tablet — one placebo oral tablet q.d.
  Arms: placebo tablets

SUMMARY:
This is a multicenter, Phase 2, double-blind, placebo-controlled study in subjects with active Ankylosing Spondylitis (AS). A total of approximately 100 subjects will be randomized to one of 2 treatment arms in a 1:1 ratio: oral filgotinib tablets q.d. or matching placebo q.d. Treatment duration will be 12 weeks. Each subject will stay in the study for a maximum of 20 weeks (from Screening visit to Follow-up visit).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects who are ≥18 years of age on the day of signing informed consent.
* Diagnosis of moderate to severe ankylosing spondylitis with documented evidence of fulfilling the Modified New York (NY) criteria
* Have active ankylosing spondylitis with a BASDAI ≥4 (numeric rating scale [NRS] 0-10) and spinal pain ≥4 (0-10 NRS) (based on BASDAI question 2, see protocol) at screening and baseline.
* Have had a documented inadequate response to NSAIDs including cyclooxygenase-2 (COX-2) inhibitors.
* If using cDMARD therapy, stable dose for at lead 4 weeks prior to Baseline.
* If using non-drug therapies (including physical therapies), these should be kept stable during screening.
* Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use highly effective methods of contraception as described in the protocol.

Key Exclusion Criteria:

* Use of JAK inhibitors, investigational or approved, at any time, including filgotinib;
* Prior use of more than one TNF inhibitor, at any time.
* Use of oral steroids at a dose >10 mg/day of prednisone or prednisone equivalent or at a dose that hasn't been stable for at least 4 weeks prior to baseline;
* Any therapy by intra-articular injections (e.g. corticosteroid, hyaluronate) within 4 weeks prior to screening;
* Use of more than 1 NSAID or COX-2 inhibitor.
* Contraindication to MRI.
* History of known or suspected complete ankylosis of the spine.
* Presence of very poor functional status or unable to perform self-care.
* Have undergone surgical treatment for ankylosing spondylitis within the last 12 weeks prior to screening.
* Administration of a live or attenuated vaccine within 12 weeks prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Ankylosing Spondylitis disease activity score (ASDAS) in filgotinib treated subjects as compared to placebo | week 12
  To evaluate the effect of filgotinib on the AS disease activity score

SECONDARY OUTCOMES:
Assessment of SpondyloArthritis international Society (ASAS) in filgotinib treated subjects as compared to placebo | week 12
  To evaluation the effect of filgotinib on the ASAS score in AS patients
Assessment by a trained joint assessor of 44 joints for tenderness (counting the number or tender joints - TJC) and swelling (counting the number of swollen joints - SJC) in filgotinib treated subjects as compared to placebo | week 12
  To evaluate the effect of filgotinib on joint tenderness and swelling in AS patient
Assessement of the Bath Ankylosing Spondylitis Disease Activity Index in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinib on BAS disease activity index in AS patients
Assessment of the Bath Ankylosing Spondylitis Functional Index in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinib on BAS functional index in AS patients
Assessment of the Bath Ankylosing Spondylitis Metrology Index in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinib on BAS metrology index in AS patients
Assessment Spondyloarthritis Research Consortium of Canada MRI in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filogtinib on Spondyloarthritis Research Consortium of Canada MRI in AS patients
Assessment of the Maastricht Ankylosing Spondylitis Enthesitis Score in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinibe on Maastricht Ankylosing Spondylitis Enthesitis Score in AS patients
Assessment of FACIT fatigue scale in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinib on FACIT fatigue scale in AS patients
Assessment of SF-36 health survey in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinib on SF-36 health survey in AS patients
Assessment of Ankylosing Spondylitis Quality of Life questionnaire (ASQoL) in filgotinib treated subjects as compared to placebo | week 12
  To assess the effect of filgotinib on ASQoL in AS patients
Difference between filgotinib treated subjects and placebo subjects in the number of Adverse events | from baseline until the final follow up visit (week 16)
  To assess safety and tolerability of filgotinib in AS patients
Difference in the number of filgotinib subjects and placebo subjects with abnormal Clinical laboratory evaluations | from baseline until the final follow up visit (week 16)
  To assess safety and tolerability of filgotinib in AS patients
Difference in the number of filgotinib treated subjects and placebo subjects with abnormal vital signs | from baseline until the final follow up visit (week 16)
  To assess safety and tolerability of filgotinib in AS patients
Difference between the number of filgotinib treated subjects and placebo subjects with abnormal physical examination | from baseline until the final follow up visit (week 16)
  To assess safety and tolerability of filgotinib in AS patients
Difference between the number of filgotinib treated subjects and placebo with abnormal ECG | At baseline, end of study visit (week 12) and final follow up visit (week 16)
  To assess safety and tolerability of filgotinib in AS patients
Difference between the number of filgotinib treated subjects and placebo with abnormal radiographic assessment | At baseline and end of study visit (week 12)
  To assess safety and tolerability of filgotinib in AS patients

CONTACTS AND LOCATIONS:
Overall Officials: Pille Harrison, MD, DPhil, MRCP (UK), Study Director — Galapagos NV
Locations (30):
- ULB Hopital Erasme, Service de Rheumatology, Brussels, Belgium
- Bulgaria (7):
  - Eurohospital, Plovdiv
  - UMHAT Kaspela EOOD, Plovdiv
  - Medical Center "Teodora", EOOD, Rousse
  - Akademik Ivan Geshov, UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - Clinic of Rheumatology, UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT "SofiaMed", OOD, Block 1, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
- Czechia (3):
  - Revmatologicka ambulance, Ostrava
  - CCBR Czech, a.s, Pardubice
  - MEDICAL PLUS s.r.o., Uherské Hradiště
- OÜ Innomedica, Tallinn, Estonia
- Poland (5):
  - Centrum Medyczne SILESIANA Sp z oo, Bytom
  - Twoja Przychodnia-Centrum Medyczne Nowa Sol, Nowa Sól
  - Ai Centrum Medyczne sp. z o.o. sp.k., Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Przychodnia Specjalistyczna, Torun
  - Centrum Medyczne AMED, Warszawa Targowek, Warsaw
- Spain (3):
  - Corporacio Sanitaria Parc Tauli, Servicio de Reumatologia, Santiago de Compostela
  - Hospital Infanta Luisa, Servicio de Reumatologia, Seville
  - Hospital Universitario Virgen Macarena, Dept. of Rheumatology, Seville
- Ukraine (10):
  - CI of Healthcare Kharkiv CCH #8 Dept of Rheumatology Kharkiv MA of PGE of MOHU, Ch of Cardiology and Funct Diagnostics, Kharkiv
  - CNI Consultative and Diagnostic Center of Pecherskyi District of Kyiv, Department of Therapy, Kiev
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Unit of Non-coronary HD&Rh, Kiev
  - CH of State Border Service of Ukraine (Military Base 2522) Dept of Therapy, D.Halytskyi Lviv NMU, Ch of Family Medicine & Dermatology, Venereology, Lviv
  - M.V. Sklifosovskyi Poltava RCH Dept of Rheumatology HSEIU UMSA, Ch of Family Medicine and Therapy, Poltava
  - CI of TRC, Ternopil
  - A.Novak Transcarpathian Regional Clinical Hospital, Dept of Rheumatology, Uzhhorod
  - M.I. Pyrogov VRCH Dept of Rheumatology M.I. Pyrogov VNMU, Ch of IM #1, Vinnytsia
  - MCIC MC LLC Health Clinic, Unit of Cardiology and Rheumatology, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Un of Therapy and CRh Dept of Therapy, Vinnytsia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maksymowych WP, Ostergaard M, Landewe R, Barchuk W, Liu K, Gilles L, Hendrikx T, Besuyen R, Baraliakos X. Filgotinib decreases both vertebral body and posterolateral spine inflammation in ankylosing spondylitis: results from the TORTUGA trial. Rheumatology (Oxford). 2022 May 30;61(6):2388-2397. doi: 10.1093/rheumatology/keab758. PMID 34647992
- [Derived] Maksymowych WP, Ostergaard M, Landewe R, Barchuk W, Liu K, Tasset C, Gilles L, Hendrikx T, Besuyen R, Baraliakos X. Impact of filgotinib on sacroiliac joint magnetic resonance imaging structural lesions at 12 weeks in patients with active ankylosing spondylitis (TORTUGA trial). Rheumatology (Oxford). 2022 May 5;61(5):2063-2071. doi: 10.1093/rheumatology/keab543. PMID 34352069
- [Derived] van der Heijde D, Baraliakos X, Gensler LS, Maksymowych WP, Tseluyko V, Nadashkevich O, Abi-Saab W, Tasset C, Meuleners L, Besuyen R, Hendrikx T, Mozaffarian N, Liu K, Greer JM, Deodhar A, Landewe R. Efficacy and safety of filgotinib, a selective Janus kinase 1 inhibitor, in patients with active ankylosing spondylitis (TORTUGA): results from a randomised, placebo-controlled, phase 2 trial. Lancet. 2018 Dec 1;392(10162):2378-2387. doi: 10.1016/S0140-6736(18)32463-2. Epub 2018 Oct 22. PMID 30360970